CLINICAL TRIAL: NCT00880178
Title: Plaque Inflammation and Dysfunctional HDL in AIM-HIGH
Acronym: HDL Proteomics
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin O'Brien, Professor of Medicine, Cardiology, University of Washington
Other Study IDs: 28201; R01HL089504 (NIH)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Atherosclerosis; Myocardial Infarction
Keywords: Simvastatin; Niacin; Vascular Disease; Magnetic Resonance Imaging; High Density Lipoprotein; Oxidation; Proteomics; Stroke; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Atherosclerosis; Myocardial Infarction; Vascular Diseases; Stroke | interventions — Simvastatin; Niacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for HDL isolation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Simvastatin: Participants in the main AIM-HIGH study who are receiving simvastatin.
  Interventions: Drug: Simvastatin
- Simvastatin and Extended-Release Niacin: Participants in the main AIM-HIGH study who are receiving simvastatin and extended-release niacin.
  Interventions: Drug: Simvastatin and Extended-Release niacin

INTERVENTIONS:
Drug: Simvastatin and Extended-Release niacin — Participants will be enrolled in this substudy only if they are candidates for the main AIM-HIGH study (NCT00120289). Participants will be randomly assigned to simvastatin or simvastatin plus niacin as a part of the main AIM-HIGH protocol, and adjustments in simvastatin and/or niacin doses will be made as per the protocol for the main AIM-HIGH study.
  Other Names: Simvastatin/Niacin
  Groups: Simvastatin and Extended-Release Niacin
Drug: Simvastatin — Participants will be enrolled in this substudy only if they are candidates for the main AIM-HIGH study (NCT00120289). Participants will be randomly assigned to simvastatin or simvastatin plus niacin as a part of the main AIM-HIGH protocol, and adjustments in simvastatin and/or niacin doses will be made as per the protocol for the main AIM-HIGH study.
  Groups: Simvastatin

SUMMARY:
Coronary heart disease (CHD) is a serious health concern that affects millions of people in the United States. It is usually caused by atherosclerosis-a condition that occurs when fatty material and plaque build up on the walls of the arteries that supply blood and oxygen to the heart, causing the arteries to narrow. As the arteries narrow, blood flow to the heart can slow down or stop, which can cause chest pain, shortness of breath, heart attack, or heart failure. Another component of CHD events involves inflammatory changes that result in structural breakdown of atherosclerotic plaques. Adding niacin to statin medications may be an effective way to block inflammation in the atherosclerotic plaques. This study will examine magnetic resonance imaging (MRI) images and blood samples of participants in the AIM-HIGH study who are taking niacin plus statins or statins alone to determine the effect of these medications on inflammation in atherosclerotic plaques.

DETAILED DESCRIPTION:
CHD is the leading cause of death in the United States. Preliminary research has shown that CHD is associated with oxidative and inflammatory changes in high-density lipoprotein (HDL) cholesterol, which is considered the "good" cholesterol. The inflammatory changes can impair HDL cholesterol's normal function, which is to remove excess cholesterol from the arteries and thereby slow the build-up of atherosclerotic plaque. Statins are cholesterol-lowering medications that are used to treat people with CHD. Taking niacin, a type of B vitamin, in combination with statins may stabilize atherosclerotic plaques better than statins alone, but more research is needed to examine how niacin may do this. By improving the ability of HDL cholesterol to repair inflammatory damage to atherosclerotic plaques, niacin may assist in preventing the inflammation that leads to plaque breakdown.

The AIM-HIGH study (NCT00120289) is examining the use of niacin plus statins in people with vascular disease. Participants in the AIM-HIGH study are randomly assigned to receive either niacin plus simvastatin, which is a type of statin medication, or simvastatin alone. The purpose of this substudy is to determine whether niacin in combination with statins reduces atherosclerotic plaque inflammation and dysfunctional HDL cholesterol more than statins alone. The substudy will enroll participants who are participating in the AIM-HIGH study. At the AIM-HIGH baseline and Year 2 study visits, study researchers for this substudy will collect an additional blood sample from participants to examine the changes in HDL oxidation levels and protein composition at both time points. Study researchers will also analyze participants' MRI scans to examine changes in plaque inflammation during the study period; these MRI scans will be completed as part of another AIM-HIGH substudy, conducted by Dr. Xue-Qiao Zhao. There will be no additional study procedures or visits for participants in this substudy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for main AIM-HIGH study (NCT00120289)
* Willing to provide informed consent for participation in this substudy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the main AIM-HIGH study (NCT00120289)
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2008-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in HDL oxidation and proteomics | Measured at Year 2

SECONDARY OUTCOMES:
Comparison of HDL oxidation and proteomics changes between participants receiving statins versus participants receiving statins plus niacin | Measured at Year 2
Comparison of change in an MRI marker of plaque inflammation between participants receiving statins versus participants receiving statins plus niacin | Measured at Year 2
Comparison of changes in HDL oxidation and proteomics with change in an MRI marker of plaque inflammation | Measured at Year 2
Change in an MRI marker of plaque inflammation | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D. O'Brien, MD, Principal Investigator — University of Washington
Locations (29):
- United States (24):
  - Cardiovascular Associates, Birmingham, Alabama
  - Cardiovascular Consultants, Phoenix, Arizona
  - Long Beach VA Medical Center, Long Beach, California
  - Christiana Care Health Services, Newark, Delaware
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - HealthPartners Riverside Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Wake Forest University, Geriatrics, Greensboro, North Carolina
  - Wake Forest University, Cardiology, Winston-Salem, North Carolina
  - Wake Forest University, Endocrinology, Winston-Salem, North Carolina
  - St. Vincent Charity Hospital, Cleveland, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Cardiology Associates, Philadelphia, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Puget Sound VA Medical Center, Seattle Campus, Seattle, Washington
- Canada (5):
  - Heart Health Institute, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Western Ontario, London, Ontario
  - St. Michael's Health Centre, Toronto, Ontario

REFERENCES:
- [Result] Chen H, Sun J, Kerwin WS, Balu N, Neradilek MB, Hippe DS, Isquith D, Xue Y, Yamada K, Peck S, Yuan C, O'Brien KD, Zhao XQ. Scan-rescan reproducibility of quantitative assessment of inflammatory carotid atherosclerotic plaque using dynamic contrast-enhanced 3T CMR in a multi-center study. J Cardiovasc Magn Reson. 2014 Aug 1;16(1):51. doi: 10.1186/s12968-014-0051-7. PMID 25084698
- [Result] Zhao XQ, Hatsukami TS, Hippe DS, Sun J, Balu N, Isquith DA, Crouse JR 3rd, Anderson T, Huston J 3rd, Polissar N, O'Brien K, Yuan C; AIM-HIGH Carotid MRI Sub-study Investigators. Clinical factors associated with high-risk carotid plaque features as assessed by magnetic resonance imaging in patients with established vascular disease (from the AIM-HIGH Study). Am J Cardiol. 2014 Nov 1;114(9):1412-9. doi: 10.1016/j.amjcard.2014.08.001. Epub 2014 Aug 13. PMID 25245415
- [Result] O'Brien KD, Hippe DS, Chen H, Neradilek MB, Probstfield JL, Peck S, Isquith DA, Canton G, Yuan C, Polissar NL, Zhao XQ, Kerwin WS. Longer duration of statin therapy is associated with decreased carotid plaque vascularity by magnetic resonance imaging. Atherosclerosis. 2016 Feb;245:74-81. doi: 10.1016/j.atherosclerosis.2015.11.032. Epub 2015 Dec 1. PMID 26708287
- [Result] O'Brien KD, Hippe DS, Chen H, Neradilek MB, Probstfield JL, Peck S, Isquith DA, Canton G, Yuan C, Polissar NL, Zhao XQ, Kerwin WS. Summary of clinical and laboratory data of study subjects with and without DCE-MRI plaque measurements in the AIM-HIGH clinical trial. Data Brief. 2016 Jan 2;6:476-81. doi: 10.1016/j.dib.2015.12.030. eCollection 2016 Mar. PMID 26977429
- [Result] Sun J, Zhao XQ, Balu N, Neradilek MB, Isquith DA, Yamada K, Canton G, Crouse JR 3rd, Anderson TJ, Huston J 3rd, O'Brien K, Hippe DS, Polissar NL, Yuan C, Hatsukami TS. Carotid Plaque Lipid Content and Fibrous Cap Status Predict Systemic CV Outcomes: The MRI Substudy in AIM-HIGH. JACC Cardiovasc Imaging. 2017 Mar;10(3):241-249. doi: 10.1016/j.jcmg.2016.06.017. PMID 28279371
- [Result] Hippe DS, Phan BAP, Sun J, Isquith DA, O'Brien KD, Crouse JR, Anderson T, Huston J, Marcovina SM, Hatsukami TS, Yuan C, Zhao XQ. Lp(a) (Lipoprotein(a)) Levels Predict Progression of Carotid Atherosclerosis in Subjects With Atherosclerotic Cardiovascular Disease on Intensive Lipid Therapy: An Analysis of the AIM-HIGH (Atherothrombosis Intervention in Metabolic Syndrome With Low HDL/High Triglycerides: Impact on Global Health Outcomes) Carotid Magnetic Resonance Imaging Substudy-Brief Report. Arterioscler Thromb Vasc Biol. 2018 Mar;38(3):673-678. doi: 10.1161/ATVBAHA.117.310368. Epub 2018 Jan 4. PMID 29301785
- [Derived] Ronsein GE, Vaisar T, Davidson WS, Bornfeldt KE, Probstfield JL, O'Brien KD, Zhao XQ, Heinecke JW. Niacin Increases Atherogenic Proteins in High-Density Lipoprotein of Statin-Treated Subjects. Arterioscler Thromb Vasc Biol. 2021 Aug;41(8):2330-2341. doi: 10.1161/ATVBAHA.121.316278. Epub 2021 Jun 17. PMID 34134520
- [Derived] Sun J, Zhao XQ, Balu N, Hippe DS, Hatsukami TS, Isquith DA, Yamada K, Neradilek MB, Canton G, Xue Y, Fleg JL, Desvigne-Nickens P, Klimas MT, Padley RJ, Vassileva MT, Wyman BT, Yuan C. Carotid magnetic resonance imaging for monitoring atherosclerotic plaque progression: a multicenter reproducibility study. Int J Cardiovasc Imaging. 2015 Jan;31(1):95-103. doi: 10.1007/s10554-014-0532-7. Epub 2014 Sep 13. PMID 25216871